CLINICAL TRIAL: NCT01352117
Title: A Randomized Evaluation of Antiretroviral Therapy Alone or With Delayed Chemotherapy Versus Antiretroviral Therapy With Immediate Adjunctive Chemotherapy for Treatment of Limited Stage AIDS-KS in Resource-Limited Settings (REACT-KS) AMC 067
Brief Title: Antiretroviral Therapy (ART) Alone or With Delayed Chemo Versus ART With Immediate Chemo for Limited AIDS-related Kaposi's Sarcoma
Acronym: REACT-KS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5264; 1U01AI068636 (NIH); AMC 067 (Other: AMC)
Record Dates: First submitted 2011-03-03; First posted 2011-05-11 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: HIV-1 Infection; Kaposi's Sarcoma
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: ART alone or with delayed ET (Active Comparator): Participants were prescribed ART (co-formulated efavirenz/emtricitabine/tenofovir disoproxil fumarate, EFV/FTC/TDF) for 96 weeks. Arm A participants who experienced KS progression on ART alone could receive ET in addition to EFV/FTC/TDF in Step 2 of the study.
  Interventions: Drug: efavirenz/emtricitabine/tenofovir disoproxil fumarate; Drug: etoposide
- Arm B: ART with immediate ET (Experimental): Participants were prescribed ART (co-formulated efavirenz/emtricitabine/tenofovir disoproxil fumarate, EFV/FTC/TDF) for 96 weeks with immediate ET for up to 16 weeks.
  Interventions: Drug: efavirenz/emtricitabine/tenofovir disoproxil fumarate; Drug: etoposide

INTERVENTIONS:
Drug: efavirenz/emtricitabine/tenofovir disoproxil fumarate — 600 mg efavirenz/200 mg emtricitabine/300 mg tenofovir disoproxil fumarate taken orally at night
  Other Names: Atripla®; EFV/FTC/TDF
Drug: etoposide — 50 mg taken orally daily from days 1-7 of each 2-week cycle. For participants without PR or CR after two cycles of therapy and no toxicity greater than Grade 2, the dose of ET was escalated to 100 mg/day orally, days 1-7, every 2 weeks. A cycle could be delayed for a maximum of 14 days. ET could not be initiated prior to 7 days after the last dose in previous cycle. ET could be administered up to a maximum of eight cycles (2 cycles during dose titration and 6 cycles at maximum dose). Participants who could not tolerate escalation of the ET dose to 100 mg/day were treated for a maximum of six cycles.
  Other Names: VePesid®; ET

SUMMARY:
AIDS-related Kaposi's sarcoma (AIDS-KS) occurs in persons with HIV infection who are also infected with the Kaposi's sarcoma herpesvirus (KSHV). Several chemotherapy (anti-cancer) drugs work well in treating KS, but there is no treatment that cures KSHV infection. One chemotherapy drug called etoposide (VePesid®, ET) has caused KS tumors to get smaller in some people.

Antiretroviral therapy (anti-HIV drugs or ART) is a group of medicines taken together to treat HIV infection. These medicines help to stop HIV from growing in the body. When this happens, the immune system, which fights infection and some cancers like KS, gets stronger. For some people, limited stage KS often improves or stays the same when they take ART. However, in some people KS continues to get worse when taking ART. These people may need chemotherapy at a later date.

This study was done to find out if taking ART with immediate etoposide (ET) is better than taking ART alone or ART with delayed ET to treat limited stage KS. The study also tried to better understand KSHV and to see what kind of side effects are caused by ART and ET and how safe ART and ET are.

DETAILED DESCRIPTION:
The study consisted of three steps. At the study Step 1 entry, the participants were randomized (1:1) to receive ART alone (Arm A) or ART with immediate ET (Arm B). Study participants in Arm A who experienced KS progression that was confirmed by the Independent Endpoint Review Committee (IERC) could receive etoposide (ET) in addition to ART by entering Step 2 between study weeks 8 and 80. The target sample size was 468, 234 per arm. Randomization was stratified by:

1. Screening CD4 cell count (<200 or ≥200 cells/mm^3) and
2. ART history (naïve or experienced).

The duration of Step 1 or Step 1 and 2 combined was 96 weeks. After 96 weeks on study, participants who received ET (Arm B participants and Arm A participants who entered Step 2) entered Step 3 for a total of 144 weeks of safety follow-up.

Step 1 visits occurred at screening, entry and weeks 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 32, 40, 48, 60, 72, 84 and 96 from study entry. Step 2 visits were scheduled at entry and weeks 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 32, 40, 48, 60, 72, 84 from Step 2 entry until up to 96 weeks on study. The key evaluations included physical examination, clinical assessments, KS exam, CD4 cell count, HIV viral load, hematology, chemistry and pregnancy testing (for women of reproductive potential). Plasma, serum, peripheral blood mononuclear cells (PBMCs), KS tumor punch biopsy were be stored for use in future analyses. Participants also completed ET and ART adherence evaluations and quality of life questionnaires. Step 3 visits were scheduled every 24 weeks and were limited to safety evaluations including targeted physical exam, clinical assessments and hematology.

Study accrual terminated early, based on the Data and Safety Monitoring Board (DSMB) recommendation in March 2016. The participants in Steps 1 and 2 at that time were arranged to enter either Step 3 for safety follow-up after ET or, if they did not receive ET, to be taken off study.

ELIGIBILITY:
Step 1: Inclusion Criteria

1. HIV-1 infection.
2. Biopsy diagnostic of KS at any time prior to study entry.
3. Limited stage KS defined as stage T0 and some presentations of stage T1. Stage T0 was confined to skin and/or lymph nodes and/or minimal oral disease defined as non-nodular KS confined to the palate. The following presentations of stage T1 KS were also eligible at the discretion of the site investigator:

   * Tumor-associated edema limited to the area(s) of KS without significant functional impairment.
   * Oral KS that consists of flat (non-nodular and non-ulcerating) lesions confined to the soft palate, hard palate, gums, and buccal mucosa.
   * Asymptomatic gastrointestinal KS (i.e., no unexplained abdominal pain or gastrointestinal bleeding).
4. A minimum of 5 cutaneous marker lesions
5. Certain laboratory values obtained within 14 days prior to study entry.
6. For female participants of reproductive potential, a negative serum or urine pregnancy test performed within 7 days prior to study entry.
7. All participants must have agreed not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization).
8. Participants who are participating in sexual activity that could lead to pregnancy must have agreed to use a combination of TWO of the following methods- Condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, IUD, tubal ligation, and/or hormone-based contraception. For Etoposide, confirmation of lack of reproductive potential was required for all participants. More information on this criterion can be found in the study protocol.
9. Ability to swallow oral medications.
10. Karnofsky performance score >= 60 within 30 days prior to entry.
11. Ability and willingness of participant or legal guardian/representative to provide informed consent.
12. Peripheral blood CD4+ lymphocyte cell count obtained within 30 days prior to study entry at a DAIDS-approved laboratory.
13. For treatment-experienced patients, the availability of an ART regimen that includes at least two ART drugs that in the opinion of the site investigator are expected to have activity based on historical genotypic testing (if available) and treatment history.
14. For participants who were to receive ART other than EFV/TDF/FTC, the availability of those ART components.

Step 2: Inclusion Criteria

1. KS progression compared to study entry or best response with ART alone while on Step 1, between weeks 8 and 80.
2. Need for ET for treatment of KS progression, in the opinion of the site investigator, after confirmation of KS progression by the IERC.
3. Willingness to receive ET for treatment of KS progression.
4. For female participants of reproductive potential, a negative serum or urine pregnancy test performed within 7 days prior to initiating ET.
5. Karnofsky Performance Score >= 50.
6. Certain laboratory values obtained within 14 days prior to Step 2 entry.
7. Ability to swallow oral medications.
8. All participants must have agreed not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization).
9. Participants who are participating in sexual activity that could lead to pregnancy must have agreed to use a combination of TWO of the following methods- Condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, IUD, tubal ligation, hormone-based contraception. For Etoposide, confirmation of lack of reproductive potential was required for all participants. More information on this criterion can be found in the study protocol.

Step 3: Inclusion Criteria

1. Received at least one dose of ET (Arm B participants and Arm A participants who entered Step 2)

Step 1: Exclusion Criteria

1. Any manifestation of KS which, in the opinion of the site investigator, requires immediate chemotherapy.
2. More than 14 days of ART after onset of KS within 6 months prior to study entry.
3. Biopsy proven KS during previous ART.
4. Breastfeeding.
5. Allergy/sensitivity to any study drug or its formulations.
6. Any prior systemic anti-neoplastic treatment for KS (including chemotherapy, biological therapy, immunotherapy or investigational therapy).
7. Any prior local treatment of cutaneous marker lesions unless there was evidence of a clear-cut progression of the lesion.
8. Receipt of any investigational therapy within 30 days prior to study entry.
9. Current or anticipated receipt of any of the prohibited medications indicated in the study protocol.
10. In the opinion of the site investigator, any psychological or social condition, or addictive disorder that would have precluded compliance with the protocol.
11. Chronic, acute, or recurrent infections that were serious, in the opinion of the site investigator, for which the participant had not completed at least 14 days of therapy prior to study entry and/or was not clinically stable.

Step 2: Exclusion Criteria

1. Chronic, acute, or recurrent infections that were serious, in the opinion of the site investigator, for which the participant had not completed at least 14 days of therapy prior to initiating ET and/or was not clinically stable.
2. Current or anticipated receipt of any of the prohibited medications indicated in the study protocol.
3. Breastfeeding.

There are no exclusion criteria for Step 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2011-11-18 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Campbell, M.D., Study Chair — University of Colorado Hospital CRS; Mina C Hosseinipour, M.D., Study Chair — University of North Carolina Lilongwe CRS
Locations (8):
- Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro, Brazil
- Walter Reed Project - Kenya Med. Research Institute Kericho CRS (12501), Kericho, Kenya
- Malawi (2):
  - College of Med. JHU CRS (30301), Blantyre
  - University of North Carolina Lilongwe CRS (12001), Lilongwe
- San Miguel CRS, San Miguel, Lima region, Peru
- South Africa (2):
  - Wits HIV CRS, Johannesburg, Gauteng
  - Durban Adult HIV CRS (11201), Durban
- JCRC CRS, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009).
- [Background] Manual for Expedited Reporting of Adverse Events to DAID, Version 2.0, January 2010. http://rsc.tech-res.com/clinical-research-sites/safety-reporting/manual
- [Background] Krown SE, Metroka C, Wernz JC. Kaposi's sarcoma in the acquired immune deficiency syndrome: a proposal for uniform evaluation, response, and staging criteria. AIDS Clinical Trials Group Oncology Committee. J Clin Oncol. 1989 Sep;7(9):1201-7. doi: 10.1200/JCO.1989.7.9.1201. PMID 2671281
- [Background] Cianfrocca M, Cooley TP, Lee JY, Rudek MA, Scadden DT, Ratner L, Pluda JM, Figg WD, Krown SE, Dezube BJ. Matrix metalloproteinase inhibitor COL-3 in the treatment of AIDS-related Kaposi's sarcoma: a phase I AIDS malignancy consortium study. J Clin Oncol. 2002 Jan 1;20(1):153-9. doi: 10.1200/JCO.2002.20.1.153. PMID 11773164
- [Result] Hosseinipour MC, Kang M, Krown SE, Bukuru A, Umbleja T, Martin JN, Orem J, Godfrey C, Hoagland B, Mwelase N, Langat D, Nyirenda M, MacRae J, Borok M, Samaneka W, Moses A, Mngqbisa R, Busakhala N, Martinez-Maza O, Ambinder R, Dittmer DP, Nokta M, Campbell TB; A5264/AMC-067 REACT-KS Team. As-Needed Vs Immediate Etoposide Chemotherapy in Combination With Antiretroviral Therapy for Mild-to-Moderate AIDS-Associated Kaposi Sarcoma in Resource-Limited Settings: A5264/AMC-067 Randomized Clinical Trial. Clin Infect Dis. 2018 Jul 2;67(2):251-260. doi: 10.1093/cid/ciy044. PMID 29365083
- [Derived] Epeldegui M, Chang D, Lee J, Magpantay LI, Borok M, Bukuru A, Busakhala N, Godfrey C, Hosseinipour MC, Kang M, Kanyama C, Langat D, Mngqibisa R, Mwelase N, Nyirenda M, Samaneka W, Hoagland B, Campbell TB, Martinez-Maza O, Krown SE; A5264/AMC-067 team. Predictive Value of Serum Biomarkers for Response of Limited-Stage AIDS-Associated Kaposi Sarcoma to Antiretroviral Therapy With or Without Concomitant Chemotherapy in Resource-Limited Settings. J Acquir Immune Defic Syndr. 2023 Oct 1;94(2):165-173. doi: 10.1097/QAI.0000000000003236. PMID 37368929
- [Derived] Kang M, Grund B, Hunsberger S, Glidden D, Volberding P. Interim monitoring in a treatment strategy trial with a composite primary endpoint. Contemp Clin Trials. 2019 Nov;86:105846. doi: 10.1016/j.cct.2019.105846. Epub 2019 Sep 11. PMID 31520741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from November 2011 to February 2016 at 10 sites in Africa and South America.
Groups:
- Arm A: ART Alone or With Delayed ET: Participants were prescribed ART for 96 weeks. Arm A participants who experienced KS progression on ART alone could receive etoposide (ET) in addition to ART in Step 2 of the study.
- Arm B: ART With Immediate ET: Participants were prescribed ART for 96 weeks with immediate etoposide (ET) for up to 16 weeks.
Period: Overall Study
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Started | 96 | 96
Entered Step 2 to Initiate Delayed ET | 32 | 0 (Only Arm A participants could enter Step 2 to receive delayed ET.)
Study Week 48 Data Potential (Enrolled >=45 weeks prior to the date when DSMB's recommendation to close the study became public.) | 80 | 83
Study Week 96 Data Potential (Enrolled >=93 weeks prior to the date when DSMB's recommendation to close the study became public.) | 58 | 61
Completed (Completed study, including the long-term safety follow-up in Step 3.) | 75 | 72
Not Completed | 21 | 24
Not completed — Death | 15 | 16
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 7
Not completed — Non-adherent to study requirements | 1 | 1
Not completed — Did not initiate study treatment | 1 | 0
Not completed — Ineligible (no KS diagnosis) | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants who initiated study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET | Total
Number analyzed (Participants) | 94 | 96 | 190
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [28 to 41] | 35 [30 to 41] | 34 [29 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 69 | 135
  Male | 28 | 27 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 83 | 86 | 169
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 30 | 32 | 62
  Brazil | 4 | 5 | 9
  Uganda | 28 | 30 | 58
  Zimbabwe | 9 | 7 | 16
  South Africa | 6 | 6 | 12
  Kenya | 15 | 13 | 28
  Peru | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 89 | 88 | 177
  White | 2 | 5 | 7
  Other | 3 | 2 | 5
HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] | 5.11 [4.48 to 5.62] | 5.10 [4.59 to 5.47] | 5.11 [4.53 to 5.50]
CD4 cell count, continuous [Median (Inter-Quartile Range); unit: cells/mm^3] | 190 [88 to 325] | 165 [63 to 327] | 184 [78 to 325]
CD4 cell count, categorized [Count of Participants; unit: Participants]
  <200 cells/mm^3 | 50 | 53 | 103
  >=200 cells/mm^3 | 44 | 43 | 87
Karnofsky score [Count of Participants; unit: Participants] — Karnofsky performance scale is from 0 (dead) to 100 (normal; no complaint; no evidence of disease) by 10.
  Participants
    60 | 1 | 0 | 1
    70 | 8 | 5 | 13
    80 | 26 | 26 | 52
    90 | 54 | 60 | 114
    100 | 5 | 5 | 10
KS stage [Count of Participants; unit: Participants] — KS tumor stage was determined by the ACTG criteria (refer to Protocol Section, References) where Stage T0 (good risk) is defined as KS confined to skin and/or lymph nodes and/or minimal oral KS and Stage T1 (poor risk) as presence of tumor-associated edema and/or presence of oral KS beyond flat lesions confined to the palate and/or presence of asymptomatic gastrointestinal KS.
  Participants
    KS tumor Stage T0 | 35 | 40 | 75
    KS tumor Stage T1 | 59 | 56 | 115
ART experience [Count of Participants; unit: Participants]
  ART-experienced | 0 | 1 | 1
  ART-naive | 94 | 95 | 189

OUTCOME MEASURES:

1. Primary Outcome: Kaposi Sarcoma (KS) Status at Week 48 Compared to Study Entry
Description: KS status is a composite, categorical outcome, ordered from worst to best as E1 (Failure: KS progression (PD), initiation of an alternate KS treatment, or no follow-up at Week 48 including death and missed visit), E2 (Stable: in follow-up at Week 48 with no KS PD nor response and without initiation of an alternate KS treatment) and E3 (Response: in follow-up at Week 48, with KS partial or complete response (PR or CR) and without initiation of an alternate KS treatment). Alternate KS treatment was defined as chemotherapy agent other than ET or other treatment triggered by worsening KS. KS outcome status (PR, stable, PR, CR) compared to study entry was evaluated at Week 48 based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). Data on initiation of alternate KS treatment, loss to follow-up and dea
Time Frame: Entry through Week 48.
Population: All eligible participants who initiated study treatment and had Study Week 48 data potential (i.e. participants enrolled at least 45 weeks prior to the date when the Data and Safety Monitoring Board's [DSMB] recommendation to close the study became public).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 80 | 83
Participants
  E1 (Failure) | 43 | 47
  E2 (Stable) | 13 | 9
  E3 (Response) | 24 | 27
Statistical Analysis 1: Comparison: Arm A: ART Alone or With Delayed ET vs Arm B: ART With Immediate ET; Test type: Superiority; p = 0.911, Wilcoxon (Mann-Whitney) — The critical value for the final analysis was adjusted for the three interim analyses conducted for the Data and Safety Monitoring Board (DSMB) review using the Haybittle-Peto guidelines, at the p-value cutoff of 0.0487; Stratified Wilcoxon-Mann-Whitney test (asymptotic method) known as van Elteren test, stratification by screening CD4 (<200 vs. >=200 cells/mm^3)

2. Secondary Outcome: KS Progressive Disease at Week 48 Compared to Study Entry
Description: KS progressive disease (PD) compared to study entry based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002).
Time Frame: Entry and Week 48
Population: All eligible participants who initiated study treatment and had Study Week 48 data potential (i.e. participants enrolled at least 45 weeks prior to the date when the DSMB's recommendation to close the study became public) who had Week 48 KS exam performed and had not initiated alternate KS treatment before Week 48.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 58 | 43
Participants
  KS PD at Week 48 | 21 | 7
  No KS PD at Week 48 | 37 | 36

3. Secondary Outcome: KS Partial Response at Week 48 Compared to Study Entry
Description: KS partial response (PR) compared to study entry based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002).
Time Frame: Entry and Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 58 | 43
Participants
  KS PR at Week 48 | 21 | 23
  No KS PR at Week 48 | 37 | 20

4. Secondary Outcome: KS Complete Response at Week 48 Compared to Study Entry
Description: KS complete response (CR) compared to study entry based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002).
Time Frame: Entry and Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 58 | 43
Participants
  KS CR at Week 48 | 3 | 4
  No KS CR at Week 48 | 55 | 39

5. Secondary Outcome: KS Partial or Complete Response at Week 48 Compared to Study Entry
Description: KS partial response (PR) or complete response (CR) compared to study entry based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002).
Time Frame: Entry and Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 58 | 43
Participants
  Week 48: KS PR or CR | 24 | 27
  Week 48: no KS PR or CR | 34 | 16

6. Secondary Outcome: Premature Study Discontinuation by Week 48
Description: Premature study discontinuation by Week 48 due to any reason, including death.
Time Frame: Entry through Week 48
Population: All eligible participants who initiated study treatment and had Study Week 48 data potential (i.e. participants enrolled at least 45 weeks prior to the date when the DSMB's recommendation to close the study became public).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 80 | 83
Participants
  Premature study discontinuation by Week 48 | 13 | 11
  No premature study discontinuation by Week 48 | 67 | 72

7. Secondary Outcome: Kaposi Sarcoma (KS) Status at Week 96 Compared to Study Entry
Description: KS status is a composite, categorical outcome, ordered from worst to best as E1 (Failure: KS PD, initiation of an alternate KS treatment, or no follow-up at Week 96 including death and missed visit), E2 (Stable: in follow-up at Week 96 with no KS progression nor response and without initiation of an alternate KS treatment) and E3 (Response: in follow-up at Week 96, with KS PR or CR and without initiation of an alternate KS treatment). Alternate KS treatment was defined as chemotherapy agent other than ET or other treatment triggered by worsening KS. KS outcome status (PD, stable, PR or CR) compared to study entry was evaluated at Week 96 based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). Data on initiation of alternate KS treatment, loss to follow-up and deaths are from entry through Week 96.
Time Frame: Entry through Week 96.
Population: All eligible participants who initiated study treatment and had Study Week 96 data potential (i.e. participants enrolled at least 93 weeks prior to the date when the DSMB's recommendation to close the study became public).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 58 | 61
Participants
  E1 (Failure) | 33 | 33
  E2 (Stable) | 4 | 0
  E3 (Response) | 21 | 28

8. Secondary Outcome: KS Progressive Disease at Week 96 Compared to Study Entry
Description: as for outcome 2
Time Frame: Entry and Week 96
Population: All eligible participants who initiated study treatment and had Study Week 96 data potential (i.e. participants enrolled at least 93 weeks prior to the date when the DSMB's recommendation to close the study became public) who had Week 96 KS exam performed and had not initiated alternate KS treatment before Week 96.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 35 | 30
Participants
  KS PD at Week 96 | 10 | 2
  No KS PD at Week 96 | 25 | 28

9. Secondary Outcome: KS Partial Response at Week 96 Compared to Study Entry
Description: as for outcome 3
Time Frame: Entry and Week 96
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 35 | 30
Participants
  KS PR at Week 96 | 19 | 24
  No KS PR at Week 96 | 16 | 6

10. Secondary Outcome: KS Complete Response at Week 96 Compared to Study Entry
Description: as for outcome 4
Time Frame: Entry and Week 96
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 35 | 30
Participants
  KS CR at Week 96 | 2 | 4
  No KS CR at Week 96 | 33 | 26

11. Secondary Outcome: KS Partial or Complete Response at Week 96 Compared to Study Entry
Description: as for outcome 5
Time Frame: Entry and Week 96
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 35 | 30
Participants
  KS PR or CR at Week 96 | 21 | 28
  No KS PR or CR at Week 96 | 14 | 2

12. Secondary Outcome: Premature Study Discontinuation by Week 96
Description: Premature study discontinuation by Week 96 due to any reason, including death.
Time Frame: Entry through Week 96
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 58 | 61
Participants
  Premature study discontinuation by Week 96 | 14 | 10
  No premature study discontinuation by Week 96 | 44 | 51

13. Secondary Outcome: Cumulative Incidence of Initial KS Progressive Disease by Week 96
Description: KS progressive disease (PD) compared to study entry or best response based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). Cumulative incidence was estimated with death and initiation of alternate KS treatment as competing risks. Time at risk was censored at the end of Step 1 (Week 96 or premature study discontinuation) or on the date when the DSMB's recommendation to close the study became public, whichever occurred earlier.
Time Frame: From entry through 96 weeks
Population: All eligible participants who initiated study treatment.
Measure: Number (95% Confidence Interval); unit: cumulative events per 100 participants
Groups:
- Arm A: ART Alone Period (Step 1): Participants were prescribed ART for 96 weeks. Arm A participants who experienced KS progression on ART alone could receive etoposide (ET) in addition to ART in Step 2 of the study. This analysis used the ART alone period (Step 1) prior to initiation of delayed ET in Step 2.
Arm/Group | Arm A: ART Alone Period (Step 1) | Arm B: ART With Immediate ET
Number analyzed (Participants) | 94 | 96
cumulative events per 100 participants | 60.61 [48.98 to 70.38] | 52.73 [40.17 to 63.82]

14. Secondary Outcome: Cumulative Incidence of Initial KS Partial or Complete Response by Week 96
Description: KS partial response (PR) or complete response (CR) compared to study entry based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). Cumulative incidence was estimated with death and initiation of delayed KS treatment (alternate KS treatment or delayed ET in Arm A) as competing risks. Time at risk was censored at the end of Step 1 (Week 96 or premature study discontinuation) or on the date when the DSMB's recommendation to close the study became public, whichever occurred earlier.
Time Frame: From entry through 96 weeks
Population: All eligible participants who initiated study treatment.
Measure: Number (95% Confidence Interval); unit: cumulative events per 100 participants
Arm/Group | Arm A: ART Alone Period (Step 1) | Arm B: ART With Immediate ET
Number analyzed (Participants) | 94 | 96
cumulative events per 100 participants | 39.89 [24.88 to 54.48] | 64.08 [51.78 to 74.01]

15. Secondary Outcome: Cumulative Incidence of Initial KS Partial Response by Week 96
Description: KS partial response (PR) compared to study entry based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). This was initially part of the outcome specified in the study protocol as "PR and CR combined and separately" to address the secondary objective on the KS response. Due to the extremely limited number of participants with KS complete response, the Statistical Analysis Plan was updated, and the Final Analysis was conducted only on the combined KS response. The outcome on PR separately was withdrawn.
Time Frame: From study treatment initiation to 96 weeks
Population: Due to the extremely limited number of participants with KS CR, KS partial response (PR) and CR were combined. The analyses of CR and PR separately which were initially specified in the study protocol were withdrawn.
Arm/Group | Arm A: ART Alone Period (Step 1) | Arm B: ART With Immediate ET
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Cumulative Incidence of Initial KS Complete Response by Week 96
Description: KS complete response (CR) compared to study entry based on clinical evaluation of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). This was initially part of the outcome specified in the study protocol as "PR and CR combined and separately" to address the secondary objective on the KS response. Due to the extremely limited number of participants with KS CR, the Statistical Analysis Plan was updated, and the Final Analysis was conducted only on the combined KS response. The outcome on CR separately was withdrawn.
Time Frame: From study treatment initiation to 96 weeks
Population: as for outcome 15
Arm/Group | Arm A: ART Alone Period (Step 1) | Arm B: ART With Immediate ET
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: Number of participants who experienced an AE (sign/symptom or laboratory abnormality) of Grade 3 or higher. The AEs were graded by the clinicians according to the Division of AIDS (DAIDS) AE Grading Table (see reference in the Protocol Section) as follows: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-Threatening.
Time Frame: From study treatment dispensation through up to Week 96, until long-term follow-up began in Step 3 or until study discontinuation.
Population: All eligible participants who initiated study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 94 | 96
Participants | 47 | 42

18. Secondary Outcome: Cumulative Incidence of KS-IRIS
Description: KS-IRIS was defined as KS progressive disease that occurs within 12 weeks of initiation of ART that is associated with an increase in peripheral blood CD4+ lymphocyte cell count of at least 50 cells/mm^3 above the study screening value and/or a decrease in the HIV RNA level by at least 0.5 log10 below the study entry value prior to, or at the time of, documented KS progressive disease. Cumulative incidence was estimated with death and initiation of alternate KS treatment as competing risks. Time at risk was censored (1) when lost to follow-up, (2) at the study visit following Week 12 or (3) on the date when the DSMB's recommendation to close the study became public, whichever occurred earlier. Time of KS-IRIS was defined as the time of the initial KS progressive disease.
Time Frame: From study entry to Week 12
Population: All eligible participants who initiated study treatment.
Measure: Number (95% Confidence Interval); unit: cumulative events per 100 participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 94 | 96
cumulative events per 100 participants | 23.14 [15.03 to 32.29] | 7.40 [3.24 to 13.85]

19. Secondary Outcome: Percentage of Participants With Etoposide Dose Modification
Description: Etoposide (ET) was administered for a maximum of 8 cycles (16 weeks) from study entry (Arm B) or from Step 2 entry (Arm A). Dose modifications were reported as temporarily held, resumed at a different dose, deferred, prematurely discontinued and underdosed. The percentage of participants who experienced each dose modification is provided in the data table below. The categories are not mutually exclusive. A participant may have experienced multiple dose modifications and may be counted in more than one category. Each participant is counted at most once within category.
Time Frame: From ET dispensation to ET discontinuation (total duration of ET was up to 16 weeks)
Population: All eligible participants who initiated study treatment. Arm A participants are limited to those who entered Step 2 to initiate delayed ET.
Measure: Number; unit: percentage of participants
Groups:
- Arm A: ART With Delayed ET (Step 2): Participants were prescribed ART for 96 weeks. Arm A participants who experienced KS progression on ART alone could receive etoposide (ET) in addition to ART in Step 2 of the study. This analysis is limited to Arm A participants who entered Step 2 to initiate delayed ET.
Arm/Group | Arm A: ART With Delayed ET (Step 2) | Arm B: ART With Immediate ET
Number analyzed (Participants) | 32 | 96
percentage of participants
  Temporarily held | 0 | 5.2
  Resumed at a different dose | 15.6 | 9.4
  Deferred | 37.5 | 24.0
  Discontinued | 6.3 | 10.4
  Underdosed | 0 | 1.0

20. Secondary Outcome: Percentage of Participants With HIV-1 RNA Suppression
Description: HIV-1 RNA suppression was defined as plasma HIV-1 RNA <400 copies/mL. Only Arm A participants could enter Step 2 to initiate delayed ET.
Time Frame: Entry and Weeks 12, 24, 32, 48, 72, 96; Step 2 entry and Weeks 12, 24, 32, 48 and 72.
Population: All eligible participants who initiated study treatment and had HIV-1 RNA results available at the specific visit. HIV-1 RNA testing was done locally using Abbott RealTime HIV-1 Test or Roche AmpliPrep/Taqman HIV-1 Test. Only Arm A participants could enter Step 2 to initiate delayed ET.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 94 | 96
percentage of participants
  Entry: HIV-1 RNA suppression | 4.3 | 4.2
  Week 12: HIV-1 RNA suppression: number analyzed (Participants) | 72 | 85
  Week 12: HIV-1 RNA suppression | 90.3 | 90.6
  Week 24: HIV-1 RNA suppression: number analyzed (Participants) | 55 | 81
  Week 24: HIV-1 RNA suppression | 94.5 | 97.5
  Week 32: HIV-1 RNA suppression: number analyzed (Participants) | 50 | 76
  Week 32: HIV-1 RNA suppression | 92.0 | 94.7
  Week 48: HIV-1 RNA suppression: number analyzed (Participants) | 43 | 72
  Week 48: HIV-1 RNA suppression | 95.3 | 98.6
  Week 72: HIV-1 RNA suppression: number analyzed (Participants) | 34 | 58
  Week 72: HIV-1 RNA suppression | 91.2 | 96.6
  Week 96: HIV-1 RNA suppression: number analyzed (Participants) | 28 | 48
  Week 96: HIV-1 RNA suppression | 92.9 | 93.8
  Step 2 entry: HIV-1 RNA suppression: number analyzed (Participants) | 30 | 0
  Step 2 entry: HIV-1 RNA suppression | 93.3 |
  Step 2 Week 12: HIV-1 RNA suppression: number analyzed (Participants) | 27 | 0
  Step 2 Week 12: HIV-1 RNA suppression | 100.0 |
  Step 2 Week 24: HIV-1 RNA suppression: number analyzed (Participants) | 24 | 0
  Step 2 Week 24: HIV-1 RNA suppression | 95.8 |
  Step 2 Week 32: HIV-1 RNA suppression: number analyzed (Participants) | 25 | 0
  Step 2 Week 32: HIV-1 RNA suppression | 96.0 |
  Step 2 Week 48: HIV-1 RNA suppression: number analyzed (Participants) | 18 | 0
  Step 2 Week 48: HIV-1 RNA suppression | 100.0 |
  Step 2 Week 72: HIV-1 RNA suppression: number analyzed (Participants) | 12 | 0
  Step 2 Week 72: HIV-1 RNA suppression | 100.0 |

21. Secondary Outcome: Percentage of Participants With ARV Dose Modification
Description: ARV dose modifications were reported as temporarily held, prematurely discontinued and increased. The percentage of participants who experienced each dose modification is provided in the data table below. The categories are not mutually exclusive. A participant may have experienced multiple dose modifications and may be counted in more than one category. Each participant is counted at most once within category.
Time Frame: From treatment dispensation to Week 96
Population: All eligible participants who initiated study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 94 | 96
percentage of participants
  Temporarily held | 7.4 | 11.5
  Prematurely discontinued | 26.6 | 21.9
  Increased | 1.1 | 0

22. Secondary Outcome: Change in log10 HIV-1 Plasma Viral Load From Entry
Description: Absolute change in log10 HIV-1 RNA from entry at study visits calculated as value at a given time point minus value at entry. This outcome was initially specified in the study protocol. However, at the first post-entry visit, most participants had unquantifiable HIV-1 RNA levels. It would be misleading to calculate change from entry to HIV RNA-1 levels that could not be quantified. Therefore, the data collected did not support the outcome and the analytic method initially proposed in the study protocol, and this outcome measure could not be analyzed. The SAP updated the HIV-1 RNA outcome measure to HIV-1 RNA suppression at study visits (please refer to the secondary outcome measure #20).
Time Frame: Entry and Weeks 12, 24, 32, 48, 72, 96; Step 2 entry and Weeks 12, 24, 32, 48 and 72.
Population: At the first post-entry visit, most participants had unquantifiable HIV-1 RNA levels. Therefore, this outcome measure could not be analyzed.
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change in Peripheral Blood CD4+ Lymphocyte Cell Count
Description: Absolute change in CD4+ cell count was calculated as value at a given visit minus the value at study screening in Step 1, and as value at a given visit minus Step 2 entry in Step 2. Only participants in Arm A could enter Step 2 to initiate delayed ET.
Time Frame: Screening and Weeks 12, 24, 32, 48, 72, 96; Step 2 entry and Weeks 12, 24, 32, 48 and 72.
Population: All eligible participants who initiated study treatment and had CD4 cell count results available at screening and the respective Step 1 visit or at Step 2 entry and the respective Step 2 visit.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
Number analyzed (Participants) | 94 | 96
cells/mm^3
  Week 12: CD4 change: number analyzed (Participants) | 71 | 85
  Week 12: CD4 change | 40 [12 to 118] | 67 [5 to 114]
  Week 24: CD4 change: number analyzed (Participants) | 55 | 82
  Week 24: CD4 change | 57 [3 to 139] | 121 [47 to 210]
  Week 32: CD4 change: number analyzed (Participants) | 49 | 76
  Week 32: CD4 change | 90 [36 to 157] | 119 [60 to 216]
  Week 48: CD4 change: number analyzed (Participants) | 43 | 72
  Week 48: CD4 change | 125 [39 to 186] | 121 [61 to 208]
  Week 72: CD4 change: number analyzed (Participants) | 34 | 58
  Week 72: CD4 change | 143 [66 to 290] | 125 [66 to 257]
  Week 96: CD4 change: number analyzed (Participants) | 28 | 47
  Week 96: CD4 change | 149 [75 to 265] | 206 [118 to 290]
  Step 2 Week 12: CD4 change: number analyzed (Participants) | 26 | 0
  Step 2 Week 12: CD4 change | -13 [-74 to 83] |
  Step 2 Week 24: CD4 change: number analyzed (Participants) | 24 | 0
  Step 2 Week 24: CD4 change | -15 [-35 to 51] |
  Step 2 Week 32: CD4 change: number analyzed (Participants) | 24 | 0
  Step 2 Week 32: CD4 change | 28 [-7 to 71] |
  Step 2 Week 48: CD4 change: number analyzed (Participants) | 17 | 0
  Step 2 Week 48: CD4 change | 2 [-108 to 143] |
  Step 2 Week 72: CD4 change: number analyzed (Participants) | 12 | 0
  Step 2 Week 72: CD4 change | 51 [-97 to 131] |

24. Secondary Outcome: Cumulative Incidence of KS Progressive Disease After Initiation of Delayed Etoposide in Arm A
Description: KS progressive disease (PD) compared to Step 2 entry (prior to initiation of delayed ET) or Step 2 best response based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). Cumulative incidence was estimated with death and initiation of alternate KS treatment as competing risks. Time at risk was censored at the end of Step 2 (at up to 84 weeks or premature study discontinuation) or on the date when the DSMB's recommendation to close the study became public, whichever occurred earlier.
Time Frame: From initiation of etoposide (Step 2 entry) to up to 84 weeks (end of Step 2)
Population: All Arm A participants who experienced KS progression and entered Step 2 to initiate delayed ET.
Measure: Number (95% Confidence Interval); unit: cumulative events per 100 participants
Groups:
- Arm A: ART With Delayed ET Period (Step 2): Participants were prescribed ART for 96 weeks. Arm A participants who experienced KS progression on ART alone could receive etoposide (ET) in addition to ART in Step 2 of the study. This analysis was limited to the ART with delayed ET period (Step 2).
Arm/Group | Arm A: ART With Delayed ET Period (Step 2)
Number analyzed (Participants) | 32
cumulative events per 100 participants | 35.78 [17.74 to 54.28]

25. Secondary Outcome: Cumulative Incidence of KS Response After Initiation of Delayed Etoposide in Arm A
Description: KS response, partial or complete (PR or CR) compared to Step 2 entry (prior to initiation of delayed ET) based on clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). Cumulative incidence was estimated with death and initiation of alternate KS treatment as competing risks. Time at risk was censored at the end of Step 2 (at up to 84 weeks or premature study discontinuation) or on the date when the DSMB's recommendation to close the study became public, whichever occurred earlier.
Time Frame: From initiation of etoposide (Step 2 entry) to up to 84 weeks (end of Step 2)
Population: All Arm A participants who experienced KS progression and entered Step 2 to initiate delayed ET.
Measure: Number (95% Confidence Interval); unit: cumulative events per 100 participants
Arm/Group | Arm A: ART With Delayed ET Period (Step 2)
Number analyzed (Participants) | 32
cumulative events per 100 participants | 62.57 [31.65 to 82.60]

ADVERSE EVENTS:
Time Frame: From study treatment dispensation to study completion at up to Week 240.
Description: The study protocol required reporting of all new diagnoses, signs/symptoms and laboratory events of >=Grade 3 and all signs/symptoms and laboratory events that led to a change in treatment, regardless of grade. All signs/symptoms and laboratory results that were observed or performed as part of establishing a diagnosis were requested regardless of grade. The DAIDS AE Grading Table (V1.0) and EAE Manual (V2.0) were used. All eligible participants who initiated study treatment are included.
Arm/Group | Arm A: ART Alone or With Delayed ET | Arm B: ART With Immediate ET
All-Cause Mortality (participants affected / at risk) | 15/94 | 16/96
Serious Adverse Events (participants affected / at risk) | 34/94 | 34/96
Other Adverse Events (participants affected / at risk) | 83/94 | 88/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: ART Alone or With Delayed ET (N=94) | Arm B: ART With Immediate ET (N=96)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 4
Bacterial sepsis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 2 | 2
Disseminated cryptococcosis (Infections and infestations) | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Hepatitis B (Infections and infestations) | 0 | 1
Malaria (Infections and infestations) | 1 | 2
Meningitis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 4
Pneumonia bacterial (Infections and infestations) | 2 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Salmonella sepsis (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 5
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hyponatraemic seizure (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: ART Alone or With Delayed ET (N=94) | Arm B: ART With Immediate ET (N=96)
Anaemia (Blood and lymphatic system disorders) | 7 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 6 | 4
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 11
Nausea (Gastrointestinal disorders) | 4 | 9
Vomiting (Gastrointestinal disorders) | 9 | 13
Chest pain (General disorders) | 9 | 10
Malaise (General disorders) | 13 | 10
Oedema peripheral (General disorders) | 14 | 4
Pain (General disorders) | 5 | 4
Peripheral swelling (General disorders) | 7 | 5
Pyrexia (General disorders) | 25 | 29
Bacteraemia (Infections and infestations) | 2 | 8
Bacterial sepsis (Infections and infestations) | 4 | 7
Malaria (Infections and infestations) | 6 | 6
Pharyngitis (Infections and infestations) | 1 | 7
Pneumonia bacterial (Infections and infestations) | 8 | 7
Pulmonary tuberculosis (Infections and infestations) | 3 | 8
Upper respiratory tract infection (Infections and infestations) | 2 | 18
Urinary tract infection (Infections and infestations) | 1 | 12
Alanine aminotransferase increased (Investigations) | 9 | 11
Aspartate aminotransferase increased (Investigations) | 14 | 18
Blood albumin decreased (Investigations) | 34 | 32
Blood alkaline phosphatase increased (Investigations) | 10 | 6
Blood bicarbonate decreased (Investigations) | 15 | 13
Blood creatinine increased (Investigations) | 4 | 6
Blood phosphorus decreased (Investigations) | 6 | 6
Blood potassium decreased (Investigations) | 3 | 5
Blood sodium decreased (Investigations) | 39 | 38
Haemoglobin decreased (Investigations) | 24 | 19
Neutrophil count decreased (Investigations) | 32 | 36
Platelet count decreased (Investigations) | 2 | 6
Weight decreased (Investigations) | 9 | 11
White blood cell count decreased (Investigations) | 6 | 7
Decreased appetite (Metabolism and nutrition disorders) | 5 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 9
Immune reconstitution inflammatory syndrome associated Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 14
Dizziness (Nervous system disorders) | 5 | 3
Headache (Nervous system disorders) | 13 | 13
Confusional state (Psychiatric disorders) | 5 | 1
Dysuria (Renal and urinary disorders) | 2 | 9
Pollakiuria (Renal and urinary disorders) | 1 | 5
Vaginal discharge (Reproductive system and breast disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 15
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less